CLINICAL TRIAL: NCT02195388
Title: Phase 1 Study - Focus On Stiffness Reduction, Endothelial Function and Autonomic Nervous System improVement in Patients After MI With or Without hypErtension After Cardiovascular Rehabilitation.
Brief Title: Focus On Stiffness Reduction, Endothelial Function and Autonomic Nervous System
Acronym: FOREVER
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Urszula Cieslik-Guerra, M.D., Medical University of Lodz
Other Study IDs: FOREVER-1
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Arterial Stiffness; Endothelial Function; Autonomic Nervous System; Acute Coronary Syndrome; Arterial Hypertension
Keywords: Arterial stiffness,; endothelial function,; autonomic nervous system,; acute coronary syndrome,; arterial hypertension,; pulse wave velocity,; augmentation index,; arterial stiffness index,; heart rate variability,; heart rate turbulence,; vascular endothelial growth factor,; asymmetric dimethylarginine
MeSH Terms: conditions — Acute Coronary Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — VEGF-A, ADMA, NT-proBNP, creatinine, uric acid, LDL, HDL, total cholesterol, trigliceride, ALT,GGTP, CRP, fibrinogen,
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CR with AH: Patients after ACS with arterial hypertension treat with comprehensive cardiac rehabilitation
  Interventions: Other: comprehensive cardiac rehabilitation
- N-CR with AH: Patients after ACS with arterial hypertension don't treat with comprehensive cardiac rehabilitation.
- CR without AH: Patients after ACS without arterial hypertension treat with comprehensive cardiac rehabilitation
  Interventions: Other: comprehensive cardiac rehabilitation

INTERVENTIONS:
Other: comprehensive cardiac rehabilitation — Standard program of comprehensive cardiac rehabilitation CR with physical activity, behavioral intervention, risk factor modification and intervention.
  Groups: CR with AH; CR without AH

SUMMARY:
Myocardial infarction is related with endothelial function, arterial stiffness and autonomic nervous system dysfunction, but also with arterial hypertension. Hypertension by itself is also related with endothelial function, arterial stiffness and autonomic nervous system dysfunction.

Primary aim of study is to investigate how complex cardiac rehabilitation influence endothelial function, arterial stiffness and autonomic nervous system activity according to presence or absence arterial hypertension.

Secondary aim is to obtain correlation between methods for the assessment of particular disorders and intercorrelation between different disorders for example endothelial function and autonomic nervous system activity.

DETAILED DESCRIPTION:
We expect that in study groups PWV will improve better that in control group. 5% of the limit value of p <0.05.

We expect that in study groups AASI will improve better that in control group. 5% of the limit value of p <0.05.

We expect that in study groups AI will improve better that in control group. 5% of the limit value of p <0.05.

We expect that time and frequency parameters of HRV will increase in study group. 5% of the limit value of p <0.05.

We expect that parameters of HRT will improve in study group. 5% of the limit value of p <0.05.

We expect improvement in RHI in study group. 5% of the limit value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* after a recent troponin-positive acute coronary syndrome (within 7-30 days) treated by means of primary coronary angioplasty,
* age 20-85 year old,
* accepted and sign informed consent,

Exclusion Criteria:

* unstable coronary artery disease,
* indications for a coronary artery bypass graft (CABG),
* peripheral artery disease,
* uncontrolled arterial hypertension,
* ventricular and supraventricular arrhythmias in excess of 10% of all the evolutions throughout the day,
* allergy to latex,
* deformities or condition after the amputation of fingers,
* body mass index (BMI) above 35 kg/m2,
* a significant hepatic or renal failure,
* infectious disease.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient after troponin-positive acute coronary syndrome (ACS) with or without arterial hypertension.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness - Pulse wave velocity (PWV) | 24 month
  Arterial stiffness will be obtained by measuring carotid-femoral pulse wave velocity using Complior device.
Arterial stiffness - Ambulatory arterial stiffness index (AASI) | 24 month
  AASI index will be calculated by non-commercial software using data from ambulatory blood pressure monitoring.
Arterial stiffness - Augmentation index (AI) | 24 month
  AI will be calculated by EndoPAT2000 system.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | 24 month
  HRV parameters in time and frequency domain will be calculated by software Cardioscan 12.
Heart rate turbulence (HRT) | 24 month
  HRT parameters will be calculated by Cardioscan 10 software.

OTHER OUTCOMES:
Endothelial function - Reactive hyperaemia index(RHI) | 24 month
  RHI parameter of microvascular endothelial function will be calculated by EndoPAT2000 system.
Endothelial function - VEGF-A, ADMA | 24 month
  Group of 40 patient will be involved in sub-study with assessment of 2 markers of endothelial function:
  Vascular Endothelial Growth Factor A (VEGF-A) will be obtained by ELISA method to assess collateral circulation development during ischemia.
  Asymmetric dimethylarginine (ADMA) will be obtained by ELISA method to assess the ability of the synthesis of nitric oxide.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Kurpesa, Professor, Study Chair — Departament of Cardiology Medical University of Lodz
Locations (1):
- Departament of Cardiology, Lodz, Łódź Voivodeship, Poland